CLINICAL TRIAL: NCT01415700
Title: Implanted Functional Electrical Stimulation of the Levators of the Ankle Versus Orthosis in the Treatment of Chronic Foot Neurological STEPPAGE-gait by Central Attack
Brief Title: Comparison Between Implanted Functional Electrical Stimulation and Foot Orthosis
Acronym: STEPSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P070155; 2007-A01444-49 (Other: ID RCB)
Record Dates: First submitted 2011-08-08; First posted 2011-08-12 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Hysterical Simulation of Disease
Keywords: feet STEPPAGE of central neurological origin; implanted functional electrical stimulation; feet orthosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stimulator (Experimental)
  Interventions: Device: Functional electrical stimulator
- Orthosis (Active Comparator)
  Interventions: Device: feet orthosis

INTERVENTIONS:
Device: Functional electrical stimulator — The stimulator is surgically implanted
  Arms: Stimulator
Device: feet orthosis — feet orthosis specifically mold
  Arms: Orthosis

SUMMARY:
The implantable feet stimulator proposes to correct the feet's STEPPAGE observed after central nervous system's injury such as hemiplegia secondary to stroke. It aims to improve the patient's walking floor by removing the STEPPAGE, reducing the effort of walking, facilitating the flow and removing anomalies compensatory (such as the mowing of the hip). Its objective is to improve the patient's autonomy locomotor.

The aim of this study is to compare the results of the implementation of an implanted stimulator in the levator muscles of the foot to the results obtained by wearing a splint-type reliever, which is considered standard treatment, in order to determine if the implanted stimulation may be proposed in the treatment of foot drop off a neurological center.

DETAILED DESCRIPTION:
The implantable feet stimulator proposes to correct the feet's STEPPAGE observed after central nervous system's injury such as hemiplegia secondary to stroke. It aims to improve the patient's walking floor by removing the STEPPAGE, reducing the effort of walking, facilitating the flow and removing anomalies compensatory (such as the mowing of the hip). Its objective is to improve the patient's autonomy locomotor.

ELIGIBILITY:
Inclusion Criteria:

* STEPPAGE foot walking in a patient with a central neurological disease
* can walk for 50 meters with or without technical assistance
* stable disease for at least 1 year
* possible walk with a brace-type reliever
* verification of possible nerve stimulation
* age greater than or equal to 18 years and under 75 years
* no toxin for 4 months
* no alcohol for 6 months
* no neurotomy for 1 year
* patient who agreed to sign an informed consent to participate in the study

Exclusion Criteria:

* cons-indication to general anesthesia
* wearing a stimulator implanted for other reasons
* patients taking neuroleptics, benzodiazepines, or antidepressants or other drugs that interfere with the quality of walking
* advanced peripheral neuropathy
* excessive restriction of passive range of ankle
* poorly controlled epilepsy
* pregnant or lactating
* non-membership of a social security scheme
* wearing orthopaedic shoes including the malleolus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Measurement of walking speed at 3 months | Measurement will be performed at 3 months
  The measurement is taken for a spontaneous march floor then fast. It follows from the establishment of the average of 3 to 5 passes on a walking track of a platform for analysis of movement
Measurement of walking speed at 6 months | Measurement will be performed at 6 months
  The measurement is taken for a spontaneous march floor then fast. It follows from the establishment of the average of 3 to 5 passes on a walking track of a platform for analysis of movement

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Decq, PUPH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France